CLINICAL TRIAL: NCT05049720
Title: ExtraVascular Implantable Cardiac Defibrillator Continued Access Study
Acronym: EV ICD CA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The NCT posting for the study has been transferred to NCT04060680
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MDT20054
Record Dates: First submitted 2021-08-26; First posted 2021-09-20 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Tachycardia; Ventricular Arrythmia
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Experimental (Experimental): Patients will be implanted with an Extravascular ICD and undergo requisite electrical testing.
  Interventions: Device: Defibrillation using the Extravascular ICD

INTERVENTIONS:
Device: Defibrillation using the Extravascular ICD — VT/VF induction attempted for defibrillation testing, as well as requisite electrical testing.

SUMMARY:
This study is designed to provide continued access to the Extravascular Implantable Cardioverter Defibrillator (EV ICD) System.

DETAILED DESCRIPTION:
The study will enroll subjects who are indicated to receive an implantable defibrillator who meet all of the inclusion criteria and none of the exclusion criteria. Subjects will receive an investigational Extravascular Implantable Cardioverter Defibrillator (EV ICD) system, in which a lead is placed outside of the heart and veins to deliver defibrillation therapy. Subjects will be followed every 6 months following system implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a Class I or IIa indication for implantation of an ICD according to the ACC/AHA/HRS Guidelines.[1]
2. Patient is willing and able to sign and date the Informed Consent Form for their participation in the study.
3. Patient is at least 18 years of age and meets age requirements per local law.
4. Patient is geographically stable and willing and able to comply with the study procedures and visits for the duration of the follow-up.

Exclusion Criteria:

1. Patient has indications for bradycardia pacing[2] or Cardiac Resynchronization Therapy (CRT)[3] (Class I, IIa, or IIb indication).
2. Patients with an existing pacemaker, ICD, or CRT device or leads.
3. Patients with these medical interventions are excluded from participation in the study:

   * Prior sternotomy
   * Any prior medical condition or procedure that leads to adhesions in the anterior mediastinal space (i.e., prior mediastinal instrumentation, mediastinitis)
   * Prior abdominal surgery in the epigastric region
   * Planned sternotomy
   * Prior chest radiotherapy

   Or any other prior/planned medical intervention not listed that precludes their participation in the opinion of the Investigator.
4. Patients with these medical conditions or anatomies are excluded from participation in the study:

   * Hiatal hernia that distorts mediastinal anatomy
   * Marked sternal abnormality (e.g., pectus excavatum that impedes the substernal tunneling path or procedure)
   * Decompensated heart failure
   * COPD with oxygen dependence
   * Gross hepatosplenomegaly

   Or any other known medical condition or anatomy type not listed that precludes their participation in the opinion of the Investigator.
5. Patients with a medical condition that precludes them from undergoing defibrillation testing:

   * Severe aortic stenosis
   * Current Intracardiac LA or LV thrombus
   * Severe proximal three-vessel or left main coronary artery disease without revascularization
   * Hemodynamic instability
   * Unstable angina
   * Recent stroke or transient ischemic attack (within the last 6 months)
   * Known inadequate external defibrillation
   * LVEF < 20%
   * LVEDD >70 mm

   Or any other known medical condition not listed that precludes their participation in the opinion of the Investigator.
6. Patient with any evidence of active infection or undergoing treatment for an infection.
7. Patient is contraindicated from temporary suspension of oral/systemic anticoagulation.
8. Patient with current implantation of neurostimulator or any other chronically implanted device that delivers current in the body.
9. Patient meets ACC/AHA/HRS or ESC clinical guideline Class III criteria for an ICD (e.g., life expectancy of less than 12 months).
10. Patient is enrolled or planning to enroll in a concurrent clinical study that may confound the results of this study, without documented pre-approval from a Medtronic study manager.
11. Patient with any exclusion criteria as required by local law (e.g., age or other).
12. Pregnant women or breastfeeding women, or women of childbearing potential and who are not on a reliable form of birth regulation method or abstinence*

(*If required by local law, women of child-bearing potential must undergo a pregnancy test within seven days prior to EV ICD Continued Access Study procedures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-07-28 (Estimated); Study Completion 2023-07-28 (Estimated)

PRIMARY OUTCOMES:
Complications | Through study completion, an average of 18 months
  EV ICD system and/or procedure related adverse events

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Khatib SM, Stevenson WG, Ackerman MJ, Bryant WJ, Callans DJ, Curtis AB, Deal BJ, Dickfeld T, Field ME, Fonarow GC, Gillis AM, Granger CB, Hammill SC, Hlatky MA, Joglar JA, Kay GN, Matlock DD, Myerburg RJ, Page RL. 2017 AHA/ACC/HRS Guideline for Management of Patients With Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2018 Oct 2;72(14):e91-e220. doi: 10.1016/j.jacc.2017.10.054. Epub 2018 Aug 16. No abstract available. PMID 29097296
- [Background] Wilkoff BL, Fauchier L, Stiles MK, Morillo CA, Al-Khatib SM, Almendral J, Aguinaga L, Berger RD, Cuesta A, Daubert JP, Dubner S, Ellenbogen KA, Mark Estes NA 3rd, Fenelon G, Garcia FC, Gasparini M, Haines DE, Healey JS, Hurtwitz JL, Keegan R, Kolb C, Kuck KH, Marinskis G, Martinelli M, McGuire M, Molina LG, Okumura K, Proclemer A, Russo AM, Singh JP, Swerdlow CD, Teo WS, Uribe W, Viskin S, Wang CC, Zhang S. 2015 HRS/EHRA/APHRS/SOLAECE expert consensus statement on optimal implantable cardioverter-defibrillator programming and testing. Heart Rhythm. 2016 Feb;13(2):e50-86. doi: 10.1016/j.hrthm.2015.11.018. Epub 2015 Dec 1. No abstract available. PMID 26607062
- [Background] Kusumoto FM, Schoenfeld MH, Barrett C, Edgerton JR, Ellenbogen KA, Gold MR, Goldschlager NF, Hamilton RM, Joglar JA, Kim RJ, Lee R, Marine JE, McLeod CJ, Oken KR, Patton KK, Pellegrini CN, Selzman KA, Thompson A, Varosy PD. 2018 ACC/AHA/HRS Guideline on the Evaluation and Management of Patients With Bradycardia and Cardiac Conduction Delay: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2019 Aug 20;74(7):e51-e156. doi: 10.1016/j.jacc.2018.10.044. Epub 2018 Nov 6. No abstract available. PMID 30412709